CLINICAL TRIAL: NCT04779918
Title: A Prospective Study Evaluating the Clinical Outcomes of Ventral or Inguinal Hernias Treated Robotically With OviTex® Reinforced Tissue Matrix
Brief Title: Ventral or Inguinal Hernia, Robotically Repaired With OviTex Mesh
Acronym: BRAVOII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tela Bio Inc (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB.2020.01.01
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hernia, Ventral; Hernia, Inguinal
Keywords: use of mesh; robotic hernia repair
MeSH Terms: conditions — Hernia, Ventral; Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OviTex Reinforced Tissue Matrix (Other): This is a single-arm study. All study subjects will receive OviTex.
  Interventions: Device: OviTex Reinforced Tissue Matrix

INTERVENTIONS:
Device: OviTex Reinforced Tissue Matrix — All study subjects will receive OviTex. All OviTex Reinforced Tissue Matrices are intended for use as a surgical mesh to reinforce or repair soft tissue where weakness exists.

SUMMARY:
This study is designed to evaluate the post-operative complications and hernia recurrence following the use of OviTex in subjects with ventral or inguinal hernias. Up to 160 subjects will participate in the study from up to 20 investigator sites.

DETAILED DESCRIPTION:
This study is intended to evaluate the post-operative complications and recurrence following the use of OviTex in ventral or inguinal hernias being treated robotically. It is a single-arm study and all subjects will receive OviTex.

ELIGIBILITY:
Inclusion Criteria:

1. Subject suffers from a ventral or inguinal hernia that requires surgical repair with the use of an implant to reinforce or replace weakened or missing tissue.
2. The patient is scheduled for an elective robotic approach with the use of OviTex LPR, OviTex Core Permanent, or OviTex 1S Permanent.
3. The size of the implant needed for repair is expected to be less than or equal to 15 x 25 cm for OviTex LPR and 25 x 40 cm for OviTex Core Permanent and OviTex 1S Permanent.
4. Subject meets CDC/SSI Wound Classification Class I (Clean), Class II (Clean-Contaminated) or Class III (Contaminated) criteria.
5. Subject is willing and able to sign an informed consent for the study and has signed the IRB approved Informed Consent form for this study.
6. Subject is able to complete Quality of Life (QoL) and pain questionnaires.
7. Subject is at least 21 years old.
8. Subject is willing to comply and able to participate fully in, and for the full duration of, the study including follow-up requirements.

Exclusion Criteria at Baseline:

1. Subject has a BMI of > 40
2. Subject meets CDC/SSI Wound Classification Class IV (Dirty-Infected) criteria
3. Subject is female and is pregnant or plans to become pregnant during the course of the study.
4. Subject has a life expectancy of < 2 years making it unlikely that the subject will successfully achieve two-year follow-up.
5. Subject has recent history of drug or alcohol abuse (in last 3 years).
6. Subject has an allergy to ovine-derived products.
7. Subject has participated in another clinical trial within the past 30 days or is currently involved in another clinical trial.
8. Subject has a strangulated hernia.

Exclusion Criteria Intraoperative:

1. Subject requires implant that cannot be introduced into the surgical site during the procedure via port or an existing incision.
2. Subject unable to receive OviTex LPR, OviTex Core Permanent, or OviTex 1S Permanent time of surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Early surgical site occurrences or wound related events | occurring within the first 3 months of the ventral or inguinal hernia repair
  Incidence of early peri- and post-operative surgical site occurrences or wound related events noted at the hernia repair site
Early post-operative complications | occurring within the first 3 months of the ventral or inguinal hernia repair.
  Incidence of other early post-operative complications

SECONDARY OUTCOMES:
Late surgical site occurrences or wound related events | occurring > 3 months after index surgery
  Incidence of late post-operative surgical site occurrences or wound related events noted at the hernia repair site
Late post-operative complications | occurring > 3 months after index surgery.
  Incidence of other late post-operative complications
Patient Reported Outcomes | Assessed at day 30, day 90, 12 months, and 24 months post-op
  Patient Reported Outcomes (QoL and pain assessments)
Hernia Recurrence | at post-operative day 90 and months 12 and 24
  True hernia recurrence at the site of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Slayden, MD, Principal Investigator — St. Lukes Hospital
Locations (10):
- United States (10):
  - University of South Alabama, Mobile, Alabama
  - SurgOne, Denver, Colorado
  - GenesisCare, Destin, Florida
  - Surgical Healing Arts Center, Fort Myers, Florida
  - St. Luke's Hospital, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - Munson Healthcare, Traverse City, Michigan
  - St. Francis Hospital, Roslyn, New York
  - Mohawk Valley Health System, Utica, New York
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No